CLINICAL TRIAL: NCT01096420
Title: Acupuncture in Chronic Migraine: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuang Tien General Hospital (Other)
Responsible Party: Principal Investigator, Chun-pai Yang, MD, Kuang Tien General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9713
Record Dates: First submitted 2010-03-29; First posted 2010-03-31 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Patients With Chronic Migraine
Keywords: chronic migraine; acupuncture; Topiramate; Randomized trial
MeSH Terms: interventions — Acupuncture Therapy; Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- acupuncture (Experimental)
  Interventions: Procedure: acupuncture
- topiramate (Active Comparator)
  Interventions: Drug: topiramate

INTERVENTIONS:
Procedure: acupuncture — Each patient had a fixed and classic acupuncture points Ex-HN-3,BL-2,GB-20,EX-HN-5 bilaterally in their 24 sessions.
  Acupuncture consisted of 24 sessions of 30 min duration, administrated over 12 weeks (two sessions per week).
  Sterile disposable and steel needle (3210) were used .
  The needles were manipulated by rotation methods to produce a characteristic sensation know as De Qi.
  Arms: acupuncture
Drug: topiramate — The patients were submitted to the topiramate treatment also for 12 consecutive weeks.
  The study phase consists of a 4-week titration and a 8-week maintenance period.
  All dosages of topiramate will be initiated at 25 mg/d hs and increased by 25 mg/d weekly to a maximum of 100 mg/day (or to the maximal tolerated dose).
  Study drug was administered daily in equally divided twice daily doses.
  Arms: topiramate

SUMMARY:
The aim of this study was to investigate the efficacy and tolerance of acupuncture treatment compared with pharmacologic treatment in patients with chronic migraines.Besides, the investigators tested whether the clinical effects of acupuncture in chronic migraine prophylaxis are mediated by changes of the plasma CGRP (Calcitonin gene-related peptide).

DETAILED DESCRIPTION:
Subjects who completed the prospective baseline periods and meet met the prespecified entry criteria will be randomized into 2 groups: acupuncture treatment, and topiramate treatment group.

Subjects will be allowed to continue taking acute migraine medications for the treatment of breakthrough attacks during the trial, but any migraine preventive medications will be prohibited.

Written informed consent was obtained from all participants before entering the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years old
* Patients were required to have a diagnosis of chronic migraine with or without medication overuse that satisfied the ICHD-2 criteria during the last 3 months prior to trial entry, with an established migraine history for at least 1 year.

Exclusion Criteria:

* Patients did not fulfill the criteria of ≧ 15 days or response to triptans or ergots on at least 8 days in prospective baseline periods .
* The presence of headaches other than chronic migraine (such as another primary chronic headache or any secondary headache).
* Migraine prophylaxis agents during last 3 months including β-blockers, anti-depressants, calcium channel blockers, anti-epileptic agents or cycle-modulating hormonal drugs.
* Migraine onset after age 50 or the age at onset of CM > 60 years.
* History of hepatic disorder, nephrolithiasis or other severe illness.
* Cognitive impairment interfering with the subject's ability to follow instructions and describe symptoms.
* Prior fearful experience of acupuncture.
* Bleeding diathesis or anticoagulation.
* Pregnant or nursing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Mean monthly number of headache days with moderate or severe intensity | 3 months
  a day with headache pain that lasts ≧ 4 h with peak severity of moderate or severe intensity, or any severity or duration if the subject takes and response to a triptan or ergot.

SECONDARY OUTCOMES:
≥ 30% or ≥ 50% reduction in mean monthly headache days with moderate or severe intensity | 3 months
Mean monthly total headache days | 3 months
Reduction from baseline in the use of acute headache medications | 3 months
Short-Form 36-Item Health Survey(SF-36) | 3 months
Beck Depression Inventory(BDI) | 3 months
Migraine disability assessment questionnaire (MIDAS) | 3 months
Plasma CGRP level | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kuang Tien General Hospital, Taichung, Taiwan, Taiwan

REFERENCES:
- [Derived] Yang CP, Chang MH, Liu PE, Li TC, Hsieh CL, Hwang KL, Chang HH. Acupuncture versus topiramate in chronic migraine prophylaxis: a randomized clinical trial. Cephalalgia. 2011 Nov;31(15):1510-21. doi: 10.1177/0333102411420585. Epub 2011 Oct 21. PMID 22019576